CLINICAL TRIAL: NCT02037321
Title: Effect of Substituting Plant Protein for Animal-Protein on Cardiometabolic Risk: A Series of Systematic Reviews and Meta-Analyses of Controlled Feeding Trials to Provide Evidence-Based Guidance for Nutrition Guidelines Development
Brief Title: Meta-Analyses of the Effect of Plant Protein Versus Animal Protein on Cardiometabolic Risk
Status: Active, not recruiting | Type: Observational
Sponsor: John Sievenpiper (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canada Research Chairs Endowment of the Federal Government of Canada (Other Government); Loblaw Companies Limited (Industry)
Responsible Party: Sponsor-Investigator, John Sievenpiper, Knowledge Synthesis Lead, University of Toronto
Organization: University of Toronto (Other)
Other Study IDs: CIHR-Plant vs animal protein
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2025-06

CONDITIONS: Diabetes; Prediabetes; Metabolic Syndrome; Dysglycemia; Overweight; Obesity; Dyslipidemia; Hypertension; Gout; Non-alcoholic Fatty Liver Disease (NAFLD); Kidney Disease; Kidney Injury; Cardiovascular Disease; Inflammation
Keywords: Systematic review and meta-analysis
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State; Metabolic Syndrome; Overweight; Obesity; Dyslipidemias; Hypertension; Gout; Non-alcoholic Fatty Liver Disease; Kidney Diseases; Cardiovascular Diseases; Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Vegetarian diets have been associated with a reduced risk of preventable diseases such as type 2 diabetes and cardiovascular disease. These effects may be mediated through direct or indirect pathways. Although the high intakes of nuts, legumes, dietary fibre, whole grains, and unsaturated plant oils have each individually been associated with lower risk of type 2 diabetes and cardiovascular disease, so too has the displacement of red meats, processed meats, and saturated animal fats. One of the most important considerations in moving from animal-based diets to more plant-based diets is the replacement of animal proteins (e.g. meat, fish, dairy, eggs) with vegetable proteins (e.g. legumes, nuts, and seeds). It is unclear whether this particular replacement alone results in advantages for metabolic and cardiovascular health. To improve evidence-based guidance for dietary guidelines and health claims development, we propose to conduct a series of systematic reviews and meta-analyses of the effect of plant-based protein in exchange for animal protein on blood lipids, glycemic control, blood pressure, body weight, uric acid, markers of non-alcoholic fatty liver disease (NAFLD), and kidney function and injury. The systematic review process allows the combining of the results from many small studies in order to arrive at a pooled estimate, similar to a weighted average, of the true effect. The investigators will be able to explore whether the effects of replacing animal-based protein for plant-based protein hold true across different sexes, age groups, and background disease states and whether the effect depends on the protein source, dose, or background diet. The findings of this proposed knowledge synthesis will help improve the health of Canadians through informing recommendations for the general public, as well as those at risk of heart disease and diabetes.

DETAILED DESCRIPTION:
Background: Vegetarian diets have been associated with a reduced risk of preventable cardiometabolic diseases such as type 2 diabetes and cardiovascular disease. It is unclear whether the replacement of animal protein with vegetable protein has cardiometabolic advantages.

Objectives: To improve evidence-based guidance for dietary guidelines and health claims development, we propose to conduct a series of systematic reviews and meta-analyses of the effects of plant-based protein in replacement for animal protein on cardiometabolic risk factors including: (1) blood lipids, (2) glycemic control, (3) blood pressure, (4) body weight, (5) uric acid, (6) markers of non-alcoholic fatty liver disease (NAFLD), (7) kidney function and injury, and (8) CRP as an inflammation marker.

Design: The planning and conduct of the proposed meta-analyses will follow the Cochrane handbook for systematic reviews of interventions. The reporting will follow the Preferred Reporting Items for Systematic reviews and Meta-Analyses (PRISMA) guidelines.

Data sources: MEDLINE, EMBASE, and The Cochrane Central Register of Controlled Trials will be searched using appropriate search terms.

Study selection: Long term (≥ 3 weeks), randomized, controlled trials that investigate the effect of exchange of plant proteins for animal proteins on the outcomes previously mentioned in humans will be included. Studies that have an acute feeding design, are not randomized, or lack a suitable control will not be included. Both isocaloric and non-isocaloric studies will be included.

Data extraction: Independent investigators (≥2) will extract information about study design, sample size, subject characteristics, pulse form, dose, follow-up, and the composition of the background diets. Mean±SEM values will be extracted for all outcomes. Standard computations and imputations will be used to derive missing variance data. Risk of bias and study quality will be assessed using the Cochrane Risk of Bias Tool and the Heyland Methodological Quality Score (MQS), respectively.

Outcomes: The proposed syntheses will each assess a set of outcomes related to a different area of cardiometabolic risk: (1) blood lipids (established therapeutic targets for the prevention of cardiovascular disease - LDL-C, apo-B, non-HDL-C), (2) glycemic control (glycated blood proteins, fasting glucose and insulin, and Homeostasis model assessment of insulin resistance [HOMA-IR]), (3) body weight, (4) uric acid, (5) blood pressure (systolic BP and diastolic BP), (6) markers of NAFLD (imaging and spectroscopy endpoints of liver fat and biomarkers of hepatocellular injury [transaminases]), (7) kidney injury and function (creatinine, urea, creatine clearance, estimated glomerular filtration rate [eGFR], albumin-to-creatine ratio [ACR], albuminuria, proteinuria) and (8) inflammation marker (CRP).

Data synthesis: Separate pooled analyses will be conducted for each area of cardiometabolic control using the Generic Inverse Variance method. Random-effects models will be used even in the absence of statistically significant between-study heterogeneity, as they yield more conservative summary effect estimates in the presence of residual heterogeneity. Exceptions will be made for the use of fixed-effects models where there is <5 included trials irrespective of heterogeneity or small trials are being pooled with larger more precise trials in the absence of statistically significant heterogeneity. Paired analyses will be applied to all crossover trials. Heterogeneity will be tested by Cochran's Q statistic and quantified by the I2 statistic. Sources of heterogeneity will be explored by sensitivity and subgroup analyses. A priori subgroup analyses will include study design, dose, vegetable protein type, animal protein comparator, follow-up, baseline values, and study quality. Significant unexplained heterogeneity will be investigated by additional post hoc subgroup analyses (e.g. age, sex, level of feeding control [metabolic, supplemented, dietary advice], washout in crossover trials, energy balance of the background diet, composition of the background diet [total % energy from fat, carbohydrate, protein], change in cholesterol intake, change in glycemic index, etc.). Meta-regression analyses will assess the significance of subgroups analyses. Publication bias will be investigated by the inspection of funnel plots and application of Egger's and Begg's tests.

Knowledge translation plan: Results will be disseminated through traditional means such as interactive presentations at local, national, and international scientific meetings and publication in high impact factor journals. Innovative means such as webcasts with e-mail feedback mechanisms will also be used. Knowledge Users will act as knowledge brokers networking among opinion leaders and different adopter groups to increase awareness at each stage. Four Knowledge Users will also participate directly as members of nutrition guidelines committees. Target adopters will include the clinical practice, public health, industry, research communities, and patient groups. Feedback will be incorporated and used to guide analyses and improve key messages at each stage.

Significance: The proposed project will demonstrate that the improvement in long term health measures. This demonstration will aid in knowledge translation related to the effects of plant proteins on cardiometabolic risk, kidney disease management, and metabolic syndrome, strengthening the evidence-base for dietary recommendations and health claims and improving health outcomes through informing healthcare providers and patients, stimulating industry innovation, and guiding future research.

ELIGIBILITY:
Inclusion Criteria:

* Dietary trials in humans
* Randomized treatment allocation
* >=3 weeks
* Suitable control (i.e. exchange with animal-protein)
* Viable endpoint data

Exclusion Criteria:

* Non-human studies
* Nonrandomized treatment allocation
* <3 weeks
* Lack of a suitable control (i.e. no exchange with animal-protein)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Varied
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2013-05; Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Glycemic control analysis | Up to 2-years
  Glycated blood proteins (HbA1c, total glycated hemoglobin, fructosamine, glycated albumin), fasting glucose, fasting insulin, and the homeostasis model assessment of insulin resistance (HOMA-IR)
Lipid control analysis | Up to 2-years
  Established therapeutic targets for cardiovascular prevention (LDL-C, apoB, non-HDL-C)
Kidney function and injury analysis | Up to 2-years
  creatinine, blood urea, creatine clearance (CrCl), estimated glomerular filtration rate (eGFR), albumin-to-creatine ratio (ACR), albuminuria, proteinuria
Body weight analysis | Up to 2-years
  body weight
Blood Pressure (BP) Analysis | Up to 2-years
  Systolic BP, diastolic BP, mean arterial pressure (MAP)
Uric acid analysis | Up to 2-years
  uric acid
Non-alcoholic fatty liver disease (NAFLD) analysis | Up to 2-years
  Imaging and spectroscopy endpoints of liver fat and biomarkers of hepatocellular injury (transaminases])
Inflammation marker, C-reactive protein (CRP) | Up to 2-years
  CRP

CONTACTS AND LOCATIONS:
Overall Officials: John L Sievenpiper, MD, PhD, Principal Investigator — Toronto 3D Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital and Department of Pathology and Molecular Medicine, Faculty of health Sciences, McMaster University; Russell J de Souza, ScD, RD, Study Director — Toronto 3D Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital and Department of Epidemiology and Biostatistics, McMaster University; Cyril WC Kendall, PhD, Study Director — Toronto 3D Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital and Department of Nutritional Sciences and Medicine, University of Toronto; David JA Jenkins, MD, PhD, DSc, Principal Investigator — Toronto 3D Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital and Department of Nutritional Sciences and Medicine, University of Toronto
Locations (1):
- Toronto 3-D (Diet, Digestive tract and Disease) Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Li SS, Blanco Mejia S, Lytvyn L, Stewart SE, Viguiliouk E, Ha V, de Souza RJ, Leiter LA, Kendall CWC, Jenkins DJA, Sievenpiper JL. Effect of Plant Protein on Blood Lipids: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Am Heart Assoc. 2017 Dec 20;6(12):e006659. doi: 10.1161/JAHA.117.006659. PMID 29263032
- [Derived] Viguiliouk E, Stewart SE, Jayalath VH, Ng AP, Mirrahimi A, de Souza RJ, Hanley AJ, Bazinet RP, Blanco Mejia S, Leiter LA, Josse RG, Kendall CW, Jenkins DJ, Sievenpiper JL. Effect of Replacing Animal Protein with Plant Protein on Glycemic Control in Diabetes: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Nutrients. 2015 Dec 1;7(12):9804-24. doi: 10.3390/nu7125509. PMID 26633472